CLINICAL TRIAL: NCT03213834
Title: Fibrinolytic Therapy Versus Medical Thoracoscopy for Treatment of Severe Pleural Infection: A Randomized Clinical Trial
Brief Title: Fibrinolytic Therapy Versus Medical Thoracoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201700012
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-09

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases | interventions — Tissue Plasminogen Activator; Deoxyribonucleases; dornase alfa

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive one of two standard-of-care treatments for severe pleural infection.
Who Masked: Outcomes Assessor
Masking Description: Change in pleural fluid volume on chest CT scan from randomization (day 0) to prior to chest tube removal will be measured by a radiologist blinded to treatment allocation using image J software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracoscopy Arm (Active Comparator): Consisting of chest thoracoscopy
  Interventions: Procedure: Chest thoracoscopy
- Fibrinolytic Therapy Arm (Active Comparator): Consisting of chest fibrinolytic therapy
  Interventions: Procedure: Chest fibrinolytic therapy; Drug: tPA; Drug: DNase

INTERVENTIONS:
Procedure: Chest thoracoscopy — Thoracoscopy will be performed as per standard protocols, with patient lateral decubitus position. Ten mLs of fluid will be collected to check for biomarkers. Adhesiolysis will be attempted and pleural irrigation will be done. At the end of the procedure, a drain will be inserted and connected to an underwater seal with a negative pressure suction
  Arms: Thoracoscopy Arm
Procedure: Chest fibrinolytic therapy — A chest tube will be inserted under ultrasonography into the most dependent area of the pleural effusion or into the largest loculation in patients with multi-loculated effusions. A of DNase and tPA will be given. Concurrent tPA and DNase will be administered intrapleurally through the chest tube followed by saline flush. The tube will then be clamped for 120 minutes and after which it will be connected back to wall suction. The intrapleural therapy will be given twice daily for a maximum of 6 doses.
  Arms: Fibrinolytic Therapy Arm
Drug: tPA — tPA administered intrapleurally through the chest tube followed by saline flush. The intrapleural therapy will be given twice daily for a maximum of 6 doses.
  Other Names: Actilyse
  Arms: Fibrinolytic Therapy Arm
Drug: DNase — DNase administered intrapleurally through the chest tube followed by saline flush. The intrapleural therapy will be given twice daily for a maximum of 6 doses.
  Other Names: pulmozyme
  Arms: Fibrinolytic Therapy Arm

SUMMARY:
The purpose of this prospective randomized clinical trial is to compare two currently accepted standard-of-care treatment strategies: medical thoracoscopy as compared to instillation of intrapleural tissue plasminogen activator (TPA) and human recombinant deoxyribonuclease (DNase) for the management of complicated pleural infections in adults as defined as complicated parapneumonic effusions or pleural empyema.

DETAILED DESCRIPTION:
Pleural infection (empyema or complex parapneumonic effusion [CPPE]) represents one of the common clinical diagnoses encountered in clinical practice in the United States (US) and worldwide. The incidence of pleural infection continues to rise with an annual incidence of approximately 65,000 in the US and United Kingdom (UK). It is associated with substantial morbidity and mortality as well as increased hospital costs despite advances in medical diagnostic and therapeutic strategies. The overall mortality of pleural infection approaches 20% and it is above 30% in elderly patients over 65 years and immunocompromised patients.

Treatment of CPPE or empyema requires antibiotics and drainage of the pleural cavity.3 However, in about 30% of cases, it is difficult to remove the fluid due to loculations, septations and increased viscosity of the pleural fluid, and around 20% will need surgical intervention to adequately treat the pleural infection.

Specific Aim 1:

To compare the efficacy of early medical thoracoscopy versus fibrinolytic therapy (tPA/DNase) in patients with complicated parapneumonic effusions or pleural empyema.

CPPE is defined as non-purulent effusion in a patient with clinical evidence of infection such as fever and/or elevated blood leukocyte count and/or elevated CRP, with pleural fluid pH ≤ 7.2 (measured by blood-gas analyzer), or pleural fluid glucose < 60 mg/dl or pleural fluid LDH >1000 IU/L26. Empyema is defined as pus within the pleural space and/or presence of bacteria on pleural fluid Gram stain or culture.

For patients to be considered for the trial they need to fulfill one of the following criteria: 1) CPPE along with evidence of septated pleural effusion on pleural ultrasonography and/or chest CT scan or 2) empyema.

ELIGIBILITY:
Inclusion Criteria:

1. CPPE along with evidence of septated pleural effusion on pleural ultrasonography and/or chest CT scan
2. empyema.

Exclusion Criteria:

1. age <18 years;
2. Pregnancy
3. inability to give informed written consent;
4. previous thoracic surgery or thrombolytic therapy for pleural infection;
5. medical thoracoscopy cannot be performed within 48 hours;
6. inability to tolerate procedure due to hemodynamic instability or severe hypoxemia;
7. inability to correct coagulopathy;
8. presence of a homogeneously echogenic effusion on pleural US27 -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiren Mehta, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kheir F, Thakore S, Mehta H, Jantz M, Parikh M, Chee A, Kaphle U, Sisnega C, Fernandez-Bussy S, Majid A. Intrapleural Fibrinolytic Therapy versus Early Medical Thoracoscopy for Treatment of Pleural Infection. Randomized Controlled Clinical Trial. Ann Am Thorac Soc. 2020 Aug;17(8):958-964. doi: 10.1513/AnnalsATS.202001-076OC. PMID 32421353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants comprised a convenience sample of adults with CPPE or empyema who presented to the UFHealth pulmonary medicine service, met all inclusion / exclusion criteria, and agreed to participate.
Pre-assignment Details: After consent, but prior to randomization, all participants underwent diagnostic thoracentesis and confirmation of pleural infection.
Period: Overall Study
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospital Days for Required to Treat Complicated Parapneumonic Effusions or Pleural Empyema.
Description: Time between initiation of treatment and hospital discharge
Time Frame: 30 days starting on day of admission
Measure: Median (Full Range); unit: days
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
days | 13 [7 to 16] | 18.5 [15 to 22]

2. Secondary Outcome: Duration of Chest Tube
Description: The number of days, during the hospital admission, where the patient demonstrated chest tube drainage
Time Frame: 30 days starting on day of admission
Measure: Median (Full Range); unit: days
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
days | 13 [6 to 13] | 7 [6 to 8]

3. Secondary Outcome: Duration of Entire Hospital Stay for Complete Treatment of Pleural Infection
Description: Number of days patient registered as in-house for treatment of pleural infection
Time Frame: 30 days starting on day of admission
Measure: Median (Full Range); unit: days
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
days | 13 [7 to 16] | 18.5 [15 to 22]

4. Secondary Outcome: Treatment Failure
Description: Following intervention, if patient requires (1) surgical intervention (VATS, open thoracotomy), (2) an additional chest tube, or (3) a repeat procedure
Time Frame: 30 days starting on day of admission
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
Participants | 2 | 1

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants who experienced documented adverse events during their hospital stays
Time Frame: 30 days starting on day of admission
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

6. Secondary Outcome: Mortality
Description: In hospital and 30 day mortality measures
Time Frame: 30 days starting on day of admission
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting at consent, and up to 12 weeks post-procedure.
Arm/Group | Thoracoscopy Arm | Fibrinolytic Therapy Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03213834/Prot_SAP_003.pdf
  • Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03213834/ICF_001.pdf